CLINICAL TRIAL: NCT01485120
Title: Accuracy Study of a Non-Invasive Forearm Blood Pressure Cuff in Comparison to an Invasive Radial Arterial Blood Pressure
Brief Title: Accuracy Study of a Non-Invasive Blood Pressure Cuff in Comparison to an Invasive Radial Arterial Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 118.02-2011-GES-0007
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Blood Pressure
Keywords: Blood pressure (low, normal, high)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Blood Pressure monitoring (Other): Blood Pressure (BP) monitoring using invasive arterial insertion as a standard reference, and an investigational, non-invasive blood pressure (NIBP) monitoring cuff. Data obtained from the cuff used the SuperSTAT NIBP algorithm and the Classic NIBP algorithm for output.
  Interventions: Device: BP monitoring using two methods

INTERVENTIONS:
Device: BP monitoring using two methods — BP readings from participant using invasive radial arterial line, Non-invasive cuff with SuperSTAT NIBP algorithm, and Non-invasive cuff with Classic NIBP algorithm.

SUMMARY:
The purpose of this study is to establish the performance of a blood pressure cuff. The hypothesis is that the blood pressure reading from the cuff will provide similar blood pressure as a radial artery.

DETAILED DESCRIPTION:
Blood pressure reading from the cuff will provide similar blood pressure as a radial artery.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent or have a legally authorized representative provide written informed consent
* Any volunteer subjects ≥ 18 years of age
* Subject must have the presence of normal sinus rhythm on ECG
* Subject will return for follow-up visit from 5 days to 8 days after study procedure

Exclusion Criteria:

* Any subject who is unable to provide written informed consent
* Any subject with the presence of peripheral vascular disease in either arm
* Any subject that demonstrates an initial NIBP screening for a blood pressure distribution range that has already been filled.
* Any subject who cannot tolerate 21 repeated BP measurements
* Any subjects with clotting or bleeding disorders
* Any subjects taking medications that are considered anticoagulants or blood thinners (For example, Clopidogrel, Warfarin, Dipyridamole, Aspirin, and Enoxaparin)
* Any subject who is unable to have arterial line placed in the radial artery
* Any subject that cannot tolerate 4 fast flushes for the frequency response
* Any female subjects pregnant or lactating
* Any subject that has previously participated in this study
* Any subjects that cannot return 5 to 8 days post study procedure for a follow-up visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ransom, MD, Principal Investigator — Clinimark, LLC
Locations (1):
- Clinimark, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Blood Pressure Monitoring: Participants with blood pressure monitored using invasive and non-invasive methods. Blood pressure monitoring will take place with both devices simultaneously. The invasive "gold standard" device is a radial arterial catheter connected to the DASH 4000, while the non-invasive device is the Soft-Cuf connected to the DASH 4000 Patient Bedside Monitor with SuperSTAT NIBP software, or same with the Classic NIBP algorithm.
Period: Overall Study
Arm/Group | Blood Pressure Monitoring
Started | 34
Completed | 32
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Blood Pressure Monitoring: Blood Pressure Monitoring using two methods: invasive radial line insertion and non-invasive blood pressure cuff
Arm/Group | Blood Pressure Monitoring
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Performance Comparison: NIBP Forearm Cuff Using SuperStat Algorithm vs. Invasive Radial Blood Pressure Reading
Description: NIBP Forearm cuff systolic and diastolic values using SuperStat algorithm compared to invasive radial blood pressure systolic and diastolic values (both obtained simultaneously).
Time Frame: Approximately 2 hours
Population: Blood Pressure (BP) monitoring using invasive arterial insertion as a standard reference, and an investigational, non-invasive blood pressure (NIBP) monitoring cuff. Data obtained from the cuff used the SuperStat algorithm for output.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Blood Pressure Monitoring: Blood Pressure (BP) monitoring using invasive arterial insertion as a standard reference, and an investigational, non-invasive blood pressure (NIBP) monitoring cuff. Data obtained from the cuff used either the SuperSTAT NIBP algorithm and the Classic NIBP algorithm for output.
Arm/Group | Blood Pressure Monitoring
Number analyzed (Participants) | 32
mmHg
  Systolic value | -0.94 (6.00)
  Diastolic value | 1.39 (3.69)

2. Primary Outcome: Performance Comparison: NIBP Forearm Cuff Using Classic Algorithm vs. Invasive Radial Blood Pressure Reading
Description: NIBP Forearm cuff systolic and diastolic values using Classic algorithm difference compared to invasive radial blood pressure readings (both readings obtained simultaneously).
Time Frame: Approximately 2 hours
Population: Blood Pressure (BP) monitoring using invasive arterial insertion as a standard reference, and an investigational, non-invasive blood pressure (NIBP) monitoring cuff. Data obtained from the cuff used the Classic NIBP algorithm for output.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Blood Pressure Monitoring: Participants with blood pressure monitored using invasive and non-invasive methods.
Arm/Group | Blood Pressure Monitoring
Number analyzed (Participants) | 32
mmHg
  Systolic value | 0.68 (7.10)
  Diastolic value | 0.42 (3.64)

ADVERSE EVENTS:
Time Frame: 2 weeks
Groups:
- Blood Pressure Monitoring: All participants enrolled in the study
Arm/Group | Blood Pressure Monitoring
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No